CLINICAL TRIAL: NCT03642860
Title: Triheptanoin's Effect on Fatty Acid Oxidation and Exercise Tolerance in Patients With Debrancher Deficiency, Glycogenin-1 Deficiency and Phosphofructoinase Deficiency at Rest and During Exercise. A Randomized, Double-blind, Placebo-controlled, Cross-over Study
Brief Title: The Effect of Triheptanoin on Fatty Acid Oxidation and Exercise Tolerance in Patients With Glycogenoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Principal Investigator, Mette Cathrine Oerngreen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #20171012 Trihep; 2017-004153-17 (EudraCT Number)
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Tarui Disease; Debrancher Deficiency; GYG1 DEFICIENCY
MeSH Terms: conditions — Glycogen Storage Disease Type VII; Glycogen Storage Disease Type III | interventions — triheptanoin; tricaprylin

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a randomized, placebo-controlled, double blind, crossover study consisting of two 14 days treatment periods set apart by minimum a 7-days wash-out period where no treatment is taken. In one treatment period, the subjects receive UX007 treatment and placebo treatment in the other. The study will consist of three separate groups; one group consisting of GSD III, one group of GSD VII, and one group of GSD XV subjects. Each of these groups will be blinded and randomized separately
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Triheptanoin oil
  Interventions: Drug: Triheptanoin
- Placebo treatment (Placebo Comparator): Safflower oil
  Interventions: Drug: Placebo Oil

INTERVENTIONS:
Drug: Triheptanoin — Daily treatment with Triheptanoin oil for 14 days (7 days titration period in addition to 7 days full dose period with 1g/kg/day).
  Other Names: Trioctanoin
  Arms: Active treatment
Drug: Placebo Oil — Daily treatment with Safflower oil for 14 days (7 days titration period in addition to 7 days full dose period with 1g/kg/day).
  Arms: Placebo treatment

SUMMARY:
The aim of this study is to investigate the effect of 14 days of treatment with the dietary oil-supplement Triheptanoin on fat metabolism and exercise tolerance in patients with Phosphofructokinase deficiency, Debrancher deficiency and Glycogenin-1 deficiency. The investigators wish to investigate whether a Triheptanoin diet can improve exercise capacity by measuring:

1. Heart rate during cycling exercise and maximal exercise capacity
2. Fat and glucose metabolism
3. Concentrations of metabolic substrates in blood during exercise
4. Perception of fatigue and symptoms by questionnaire
5. Degree of exhaustion during cycling exercise by Borg score

All measurements are done before and after 14 days with a Triheptanoin-oil diet, and before and after 14 days diet with safflower (Placebo-oil).

Triheptanoin-oil supplementation in the diet has been shown to increase metabolism of both fat and carbohydrates in patients with other metabolic myopathies. In these patients, Triheptanoin improved physical performance and has reduced the amount of symptoms experienced by patients.

DETAILED DESCRIPTION:
BACKGROUND:

Neuromuscular diseases affect more than 5% of the population in Western countries. Some of the more rare neuromuscular disorders are patients with metabolic myopathies, which are hereditary disorders caused by enzymatic defects of intermediary metabolism. The disorders are generally subdivided in two major groups affecting either carbohydrate metabolism (the glycogenosis) or lipid metabolism. Patients suffer from recurrent episodes of exercise intolerance, muscle pain and muscle contractures/stiffness, and in severe cases rhabdomyolysis (breakdown of skeletal muscle fibers) and myoglobinuria. Recognition of the metabolic block in the metabolic myopathies has started the development of new therapeutic options. Enzyme replacement therapy with recombinant lysosomal acid alpha-glucosidase (rGAA) has revolutionized treatment of early onset Pompe's disease, glycogen storage disease (GSD) II.(1-3) Supplements of riboflavin, carnitine and sucrose show promise in patients with respectively riboflavin-responsive multiple acyl-Coenzyme A (CoA) dehydrogenase deficiency (4), primary carnitine deficiency (5-7) and McArdle disease (8). However, for many of the glycogenosis treatment primarily relies on avoiding precipitating factors, and dietary supplements that bypass the metabolic block.(9) Only a few of the used supplements are validated, and further studies are needed to define efficacious treatments.

A promising product for treatment of glycogenosis is Triheptanoin. Triheptanoin provides patients with medium-length, odd-chain fatty acids that are metabolized into ketones, which replace deficient intermediates in the Tricaboxylic acid (TCA) cycle, thus supporting glucose production through gluconeogenesis, resulting in a lower turnover of glycogen.(10) Triheptanoin has primarily been used in lipid metabolism disorders, where it has shown a remarkable improvement of cardiac and muscular symptoms in three children with VLCAD deficiency and in seven patients with Carnitine palmitoyltransferase (CPT) II deficiency after dietary Triheptanoin supplementation.(10,11)

Metabolic studies in patients with the glycogenosis McArdle disease and Debrancher deficiency has showed that these disorders are associated with an energy deficit caused by reduced skeletal muscle oxidation of carbohydrates and a compensatory increase in fatty acid oxidation. Despite increasing availability of free fatty acid (FFA) during exercise, fatty acid oxidation (FAO) is not increased further, even though the energy deficit is maintained.(12,13)

McArdle disease is one of the largest and most investigated groups of the muscle glycogenosis, caused by mutations in the myophosphorylase gene (PYGM) on chromosome 11 that encodes muscle glycogen phosphorylase.(14). It is know that TCA cycle intermediates are low during exercise in patients with McArdle disease, and most likely the impaired FAO relates to a slowing of the TCA-cycle by limited supply from glycolysis.(15) Triheptanoin, most likely can correct the suspected shortage of anaplerotic intermediates to spark the TCA-cycle in patients with glycogenosis as well, and studies are ongoing in patients with McArdle disease at our research unit Copenhagen Neuromuscular Center. Clinical-Trials.gov Identifier: NCT02432768.

Other glycogenoses as Debrancher deficiency, Phosphofructokinase deficiency and Glycogenin 1 deficiency, all involved in either glycogenolysis or gluconeogenesis might benefit from Triheptanoin treatment.

Glycogen storage disease III (GSD III) also known as Debrancher deficiency or Cori-Forbes disease is caused by deficient activity of glycogen debranching enzyme (GDE) due to mutations in the AGL gene on chromosome 1p21. (16) More than 20 different disease-causing mutations have been identified in this gene.(17) Debranching enzyme is required for complete hydrolysis of glycogen and GSD III is associated with an accumulation of abnormal glycogen with short outer chains.(18) Four subtypes are described:

1. Type IIIa (the most common) that affects enzymes in the liver and the skeletal and cardiac muscle.
2. Type IIIb (about 15% of patients) involves only the liver enzyme.
3. Type IIIc (rare) with a selective loss of only one of the two GDE activities affecting muscle.
4. Type IIId (rare) with loss of the transferase affecting muscle and liver (19) Dominant features during infancy and childhood are hepatomegaly, hypoglycaemia, hyperlipidaemia, and growth retardation.(16) Muscle weakness (myopathy) and wasting typically present in the third decade. Weakness can be both proximal and distal. Electromyography (EMG) and muscle histology show myopathic changes and large glycogen deposits in the muscle.(20) Treatment is symptomatic. GSD III is associated with fixed skeletal muscle weakness and some patients have exercise-related dynamic symptoms, most likely caused by a reduced skeletal muscle oxidation of carbohydrates and a compensatory increase in fatty acid oxidation.(13,21) Phosphofructokinase deficiency (GSD VII) is another glycogenosis inherited in an autosomal recessive manner causing a defect in the rate-limiting enzyme of glycolysis, phosphofructokinase (PFK).(22) The defect results in a complete block in muscle glycolysis and glycogenolysis. Clinical features are exercise intolerance, myopathy and muscle contractures that can lead to myoglobinuria. The exercise intolerance is due to a severely restricted oxidative metabolism. An increase in blood glucose will actually decrease exercise tolerance in GSD VII contrary to GSD IIIa where it has an increasing effect. Therefore, the GSD VII subjects depend on the availability of blood borne fuels such as free fatty acids and ketones seen during fasting. (23) Glycogenin-1(GYG1) deficiency (GSD XV) (OMIM #613507) is an inborn error of glycogen synthesis caused by mutations in the GYG1 gene. GYG1 works as the initial building block in the biosynthesis of glycogen in skeletal muscle. It is a glycosyl-transferase that uses UDP-glucose as substrate for autoglycosylation, forming an oligosaccharide by the process of UDP-alpha-D-glucose + glycogenin -> UDP + alpha-D-glucosylglycogenin.(24) GYG1 deficiency is inherited autosomal recessively, and is the most recently discovered muscle glycogenosis.

Most patients present with a slowly progressive adult-onset myopathy with a variable clinical presentation.(25) Some adult patients also report exercise intolerance.(26-28) Metabolic studies show that patients with GYG1 deficiency, not only have abnormal formation of glycogen, but also have impaired muscle glycogenolysis, as suggested by impaired lactate production during exercise and improved exercise tolerance with glucose infusion; results are accepted for publication in Neurology.

At present, there is only 1 known patient with Debrancher deficiency, no patients with PFK deficiency and two patients with GYG1 deficiency in Denmark. Therefore the study will aim to include patients from abroad. Patients will fly in for studies in Copenhagen, as the investigators have done many times before.(12,29-31)

Based on observation from Roe et al. and Mochel et al. the first effects of Triheptanoin appears within 48 hrs of treatment. Furthermore, based on these observations the treatment period will consist of a week of dosage escalation to avoid potential gastro-intestinal side effects.(10,11,32-34) Therefore, the investigators hypothesize that 14 days of treatment with Triheptanoin oil will improve exercise tolerance, indicated by heart rate, and fatty acid oxidation during steady state cycling exercise using indirect calorimetry and stable isotope technique in patients with the glycogenosis Debrancher deficiency, PFK deficiency and GYG1 deficiency.

INVESTIGATIONAL PRODUCT:

UX007 (Triheptanoin) is an artificially made oil of a triglyceride of three 7-carbon fatty acid chains (heptanoate) that can be used in the treatment of patients with several types of inborn errors of metabolism associated with an impaired functioning of the TCA.(10,11,32-34)(See Investigator's Brochure). UX007 (Triheptanoin) is a liquid, intended for PO administration. UX007 is a colorless to yellow oil supplied in 1 L round amber-colored glass bottles. UX007 is manufactured, packaged, and labeled according to Good Manufacturing Procedure (GMP) regulations.

Processes that replenish the stores of TCA-intermediates are called anaplerosis. Metabolism of odd-numbered carbon fatty acids such as Triheptanoin provides anaplerotic substrates through ketone body production in the liver and beta-oxidation in peripheral tissues, which forms propionyl- and acetyl-CoA that both enter the TCA-cycle.(32-35) The effect of the UX007-intake will be compared to intake of a placebo substance. Placebo will consist of safflower oil and will match the appearance of UX007, which is orally administered in the same manner as UX007.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age >15 years
* Genetically and/or biochemically verified diagnosis of Debrancher deficiency or Phosphofructokinase deficiency or Glycogenin 1 deficiency
* Capacity to consent
* All women in fertile age must be on contraceptive treatment with: Birth control pills, coil, ring, transdermal hormone patch injection of synthetic progesterone or subdermal implant.

Exclusion Criteria:

* Significant cardiac or pulmonary disease
* Pregnancy (confirmed by urine stick) or breastfeeding.
* Treatment with beta-blockers
* Inability to perform cycling exercise
* Any other significant disorder that may confound the interpretation of the findings.
* Subjects at risk of musculoskeletal injury, i.e. with disease in joints or muscle.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Heart rate | 60 min
  Heart rate during constant load cycling exercise.
Palmitate oxidation | 60 min
  Palmitate oxidation measured via stable isotope technique and indiret calorimetry during constant load exercise.

SECONDARY OUTCOMES:
Short Form-36 Questionnaire | 2 weeks
  The Short form-36 assesses eight health concepts: limitations in Quality of life physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems); bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. The standard form of the instruments asks for participants to reply to questions according to how they have felt over the previous week. The items use Likert-type scales, from 1-5 points, where 1 usually indicates that the patient is feeling worse.
Maximal workload capacity | 60 min
  During cycle exercise
Plasma concentrations of lactate, ammonia, glucose, FFA, acyl-carnitines, malate, C5, insulin, adrenalin and noradrenalin. | 60 min
Rate of Perceived Exertion (RPE) | 60 min
  Borg Score during constant workload cycling. The Borg RPE scale is a numerical scale that ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion. The Borg scale is named after Borg GA 1982.
Bouchards energy expenditure questionnaire | 3 days
  Bouchard's Physical Activity Record (BAR) is a widely used diary in which participants report physical activity for each 15 minute interval over three days. Activities are rated on a scale of 1 to 9 (1 = sedentary activity, 9 = intense manual work or high intensity sports) to yield a total energy expenditure score.
Glucose rate of appearance and disappearance | 60 min

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harris, R. & Devlin, T. Textbook of Biochemistry with Clinical Correlations. 1997, (Wiley-Liss).
- [Result] van der Ploeg AT, Barohn R, Carlson L, Charrow J, Clemens PR, Hopkin RJ, Kishnani PS, Laforet P, Morgan C, Nations S, Pestronk A, Plotkin H, Rosenbloom BE, Sims KB, Tsao E. Open-label extension study following the Late-Onset Treatment Study (LOTS) of alglucosidase alfa. Mol Genet Metab. 2012 Nov;107(3):456-61. doi: 10.1016/j.ymgme.2012.09.015. Epub 2012 Sep 17. PMID 23031366
- [Result] van der Ploeg AT, Clemens PR, Corzo D, Escolar DM, Florence J, Groeneveld GJ, Herson S, Kishnani PS, Laforet P, Lake SL, Lange DJ, Leshner RT, Mayhew JE, Morgan C, Nozaki K, Park DJ, Pestronk A, Rosenbloom B, Skrinar A, van Capelle CI, van der Beek NA, Wasserstein M, Zivkovic SA. A randomized study of alglucosidase alfa in late-onset Pompe's disease. N Engl J Med. 2010 Apr 15;362(15):1396-406. doi: 10.1056/NEJMoa0909859. PMID 20393176
- [Result] van der Ploeg AT, Reuser AJ. Pompe's disease. Lancet. 2008 Oct 11;372(9646):1342-53. doi: 10.1016/S0140-6736(08)61555-X. PMID 18929906
- [Result] Olsen RK, Olpin SE, Andresen BS, Miedzybrodzka ZH, Pourfarzam M, Merinero B, Frerman FE, Beresford MW, Dean JC, Cornelius N, Andersen O, Oldfors A, Holme E, Gregersen N, Turnbull DM, Morris AA. ETFDH mutations as a major cause of riboflavin-responsive multiple acyl-CoA dehydrogenation deficiency. Brain. 2007 Aug;130(Pt 8):2045-54. doi: 10.1093/brain/awm135. Epub 2007 Jun 20. PMID 17584774
- [Result] Longo N, Amat di San Filippo C, Pasquali M. Disorders of carnitine transport and the carnitine cycle. Am J Med Genet C Semin Med Genet. 2006 May 15;142C(2):77-85. doi: 10.1002/ajmg.c.30087. PMID 16602102
- [Result] Scholte HR, Rodrigues Pereira R, de Jonge PC, Luyt-Houwen IE, Hedwig M, Verduin M, Ross JD. Primary carnitine deficiency. J Clin Chem Clin Biochem. 1990 May;28(5):351-7. PMID 2199596
- [Result] Lamhonwah AM, Olpin SE, Pollitt RJ, Vianey-Saban C, Divry P, Guffon N, Besley GT, Onizuka R, De Meirleir LJ, Cvitanovic-Sojat L, Baric I, Dionisi-Vici C, Fumic K, Maradin M, Tein I. Novel OCTN2 mutations: no genotype-phenotype correlations: early carnitine therapy prevents cardiomyopathy. Am J Med Genet. 2002 Aug 15;111(3):271-84. doi: 10.1002/ajmg.10585. PMID 12210323
- [Result] Andersen ST, Haller RG, Vissing J. Effect of oral sucrose shortly before exercise on work capacity in McArdle disease. Arch Neurol. 2008 Jun;65(6):786-9. doi: 10.1001/archneur.65.6.786. PMID 18541798
- [Result] Orngreen MC, Vissing J. Treatment Opportunities in Patients With Metabolic Myopathies. Curr Treat Options Neurol. 2017 Sep 21;19(11):37. doi: 10.1007/s11940-017-0473-2. PMID 28932990
- [Result] Roe CR, Yang BZ, Brunengraber H, Roe DS, Wallace M, Garritson BK. Carnitine palmitoyltransferase II deficiency: successful anaplerotic diet therapy. Neurology. 2008 Jul 22;71(4):260-4. doi: 10.1212/01.wnl.0000318283.42961.e9. PMID 18645163
- [Result] Roe CR, Sweetman L, Roe DS, David F, Brunengraber H. Treatment of cardiomyopathy and rhabdomyolysis in long-chain fat oxidation disorders using an anaplerotic odd-chain triglyceride. J Clin Invest. 2002 Jul;110(2):259-69. doi: 10.1172/JCI15311. PMID 12122118
- [Result] Orngreen MC, Jeppesen TD, Andersen ST, Taivassalo T, Hauerslev S, Preisler N, Haller RG, van Hall G, Vissing J. Fat metabolism during exercise in patients with McArdle disease. Neurology. 2009 Feb 24;72(8):718-24. doi: 10.1212/01.wnl.0000343002.74480.e4. PMID 19237700
- [Result] Preisler N, Laforet P, Madsen KL, Prahm KP, Hedermann G, Vissing CR, Galbo H, Vissing J. Skeletal muscle metabolism is impaired during exercise in glycogen storage disease type III. Neurology. 2015 Apr 28;84(17):1767-71. doi: 10.1212/WNL.0000000000001518. Epub 2015 Apr 1. PMID 25832663
- [Result] Burke J, Hwang P, Anderson L, Lebo R, Gorin F, Fletterick R. Intron/exon structure of the human gene for the muscle isozyme of glycogen phosphorylase. Proteins. 1987;2(3):177-87. doi: 10.1002/prot.340020303. PMID 3447177
- [Result] Sahlin K, Jorfeldt L, Henriksson KG, Lewis SF, Haller RG. Tricarboxylic acid cycle intermediates during incremental exercise in healthy subjects and in patients with McArdle's disease. Clin Sci (Lond). 1995 Jun;88(6):687-93. doi: 10.1042/cs0880687. PMID 7634753
- [Result] Coleman RA, Winter HS, Wolf B, Gilchrist JM, Chen YT. Glycogen storage disease type III (glycogen debranching enzyme deficiency): correlation of biochemical defects with myopathy and cardiomyopathy. Ann Intern Med. 1992 Jun 1;116(11):896-900. doi: 10.7326/0003-4819-116-11-896. PMID 1580445
- [Result] Shen J, Bao Y, Liu HM, Lee P, Leonard JV, Chen YT. Mutations in exon 3 of the glycogen debranching enzyme gene are associated with glycogen storage disease type III that is differentially expressed in liver and muscle. J Clin Invest. 1996 Jul 15;98(2):352-7. doi: 10.1172/JCI118799. PMID 8755644
- [Result] Van Hoof F, Hers HG. The subgroups of type 3 glycogenosis. Eur J Biochem. 1967 Oct;2(3):265-70. doi: 10.1111/j.1432-1033.1967.tb00134.x. No abstract available. PMID 5235982
- [Result] Ding JH, de Barsy T, Brown BI, Coleman RA, Chen YT. Immunoblot analyses of glycogen debranching enzyme in different subtypes of glycogen storage disease type III. J Pediatr. 1990 Jan;116(1):95-100. doi: 10.1016/s0022-3476(05)81652-x. PMID 2295969
- [Result] Kishnani PS, Austin SL, Arn P, Bali DS, Boney A, Case LE, Chung WK, Desai DM, El-Gharbawy A, Haller R, Smit GP, Smith AD, Hobson-Webb LD, Wechsler SB, Weinstein DA, Watson MS; ACMG. Glycogen storage disease type III diagnosis and management guidelines. Genet Med. 2010 Jul;12(7):446-63. doi: 10.1097/GIM.0b013e3181e655b6. PMID 20631546
- [Result] Preisler N, Pradel A, Husu E, Madsen KL, Becquemin MH, Mollet A, Labrune P, Petit F, Hogrel JY, Jardel C, Maillot F, Vissing J, Laforet P. Exercise intolerance in Glycogen Storage Disease Type III: weakness or energy deficiency? Mol Genet Metab. 2013 May;109(1):14-20. doi: 10.1016/j.ymgme.2013.02.008. Epub 2013 Feb 19. PMID 23507172
- [Result] Haller RG, Lewis SF. Glucose-induced exertional fatigue in muscle phosphofructokinase deficiency. N Engl J Med. 1991 Feb 7;324(6):364-9. doi: 10.1056/NEJM199102073240603. PMID 1824792
- [Result] Viskupic E, Cao Y, Zhang W, Cheng C, DePaoli-Roach AA, Roach PJ. Rabbit skeletal muscle glycogenin. Molecular cloning and production of fully functional protein in Escherichia coli. J Biol Chem. 1992 Dec 25;267(36):25759-63. PMID 1281472
- [Result] Moslemi AR, Lindberg C, Nilsson J, Tajsharghi H, Andersson B, Oldfors A. Glycogenin-1 deficiency and inactivated priming of glycogen synthesis. N Engl J Med. 2010 Apr 1;362(13):1203-10. doi: 10.1056/NEJMoa0900661. PMID 20357282
- [Result] Malfatti E, Nilsson J, Hedberg-Oldfors C, Hernandez-Lain A, Michel F, Dominguez-Gonzalez C, Viennet G, Akman HO, Kornblum C, Van den Bergh P, Romero NB, Engel AG, DiMauro S, Oldfors A. A new muscle glycogen storage disease associated with glycogenin-1 deficiency. Ann Neurol. 2014 Dec;76(6):891-8. doi: 10.1002/ana.24284. Epub 2014 Oct 31. PMID 25272951
- [Result] Akman HO, Aykit Y, Amuk OC, Malfatti E, Romero NB, Maioli MA, Piras R, DiMauro S, Marrosu G. Late-onset polyglucosan body myopathy in five patients with a homozygous mutation in GYG1. Neuromuscul Disord. 2016 Jan;26(1):16-20. doi: 10.1016/j.nmd.2015.10.012. Epub 2015 Nov 10. PMID 26652229
- [Result] Luo S, Zhu W, Yue D, Lin J, Wang Y, Zhu Z, Qiu W, Lu J, Hedberg-Oldfors C, Oldfors A, Zhao C. Muscle pathology and whole-body MRI in a polyglucosan myopathy associated with a novel glycogenin-1 mutation. Neuromuscul Disord. 2015 Oct;25(10):780-5. doi: 10.1016/j.nmd.2015.07.007. Epub 2015 Jul 15. PMID 26255073
- [Result] Orngreen MC, Madsen KL, Preisler N, Andersen G, Vissing J, Laforet P. Bezafibrate in skeletal muscle fatty acid oxidation disorders: a randomized clinical trial. Neurology. 2014 Feb 18;82(7):607-13. doi: 10.1212/WNL.0000000000000118. Epub 2014 Jan 22. PMID 24453079
- [Result] ORngreen MC, Norgaard MG, Sacchetti M, van Engelen BG, Vissing J. Fuel utilization in patients with very long-chain acyl-coa dehydrogenase deficiency. Ann Neurol. 2004 Aug;56(2):279-83. doi: 10.1002/ana.20168. PMID 15293280
- [Result] Orngreen MC, Schelhaas HJ, Jeppesen TD, Akman HO, Wevers RA, Andersen ST, ter Laak HJ, van Diggelen OP, DiMauro S, Vissing J. Is muscle glycogenolysis impaired in X-linked phosphorylase b kinase deficiency? Neurology. 2008 May 13;70(20):1876-82. doi: 10.1212/01.wnl.0000289190.66955.67. Epub 2008 Apr 9. PMID 18401027
- [Result] Roe CR, Mochel F. Anaplerotic diet therapy in inherited metabolic disease: therapeutic potential. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):332-40. doi: 10.1007/s10545-006-0290-3. PMID 16763896
- [Result] Mochel F, DeLonlay P, Touati G, Brunengraber H, Kinman RP, Rabier D, Roe CR, Saudubray JM. Pyruvate carboxylase deficiency: clinical and biochemical response to anaplerotic diet therapy. Mol Genet Metab. 2005 Apr;84(4):305-12. doi: 10.1016/j.ymgme.2004.09.007. PMID 15781190
- [Result] Roe CR, Bottiglieri T, Wallace M, Arning E, Martin A. Adult Polyglucosan Body Disease (APBD): Anaplerotic diet therapy (Triheptanoin) and demonstration of defective methylation pathways. Mol Genet Metab. 2010 Oct-Nov;101(2-3):246-52. doi: 10.1016/j.ymgme.2010.06.017. Epub 2010 Jul 6. PMID 20655781
- [Result] Brunengraber H, Roe CR. Anaplerotic molecules: current and future. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):327-31. doi: 10.1007/s10545-006-0320-1. PMID 16763895